CLINICAL TRIAL: NCT06700382
Title: A Cohort Study of Different Methods of Adjuvant Capecitabine Regimens in Patients With Non-PCR After Neoadjuvant Therapy for Triple Negative Breast Cancer
Brief Title: Different Methods of Capecitabine in Patients With Non-PCR After Neoadjuvant Therapy for TNBC
Acronym: NeoTNBCX
Status: Recruiting | Type: Observational
Sponsor: Shu Wang (Other)
Responsible Party: Sponsor-Investigator, Shu Wang, director of breast center, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: PKUPH2024Z167
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Triple Negative Breast Cancer
Keywords: neoadjuvant chemotherapy; adjuvant chemotherapy; non-pCR; capecitabine
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6-8 cycles full dose capecitabine: 6-8 cycles of full dose capecitabine intensive therapy (1250mg/m2, BID,D1-D14,Q3W)
  Interventions: Drug: capecitabine
- 1-year metronomic capecitabine: 1-year capecitabine metronomic chemotherapy (650mg/m2,BID)
  Interventions: Drug: capecitabine
- no other chemotherapy: no other chemotherapy besides neoadjuvant therapy

INTERVENTIONS:
Drug: capecitabine — different methods of treatment for capecitabine
  Groups: 1-year metronomic capecitabine; 6-8 cycles full dose capecitabine

SUMMARY:
The survival rate of patients with pathological complete response (pCR) after neoadjuvant therapy was significantly better than that of patients with tumor residue, that is, non-pCR patients. Therefore, studies have confirmed that intensive adjuvant therapy for patients with non-pCR after neoadjuvant chemotherapy can further improve the survival of this population. Previous studies have given capecitabine treatment to such patients as standard. However, it is unknown whether capecitabine intensification still has the same status under the premise that most patients receive immunotherapy at the neoadjuvant stage; Whether there are differences in the efficacy and safety of capecitabine standard 6-8 cycle intensive regimen and capecitabine metronomic chemotherapy are practical problems encountered in clinical practice. This study explored the efficacy and safety of 6-8 cycles of full dose capecitabine intensive therapy compared with 1-year capecitabine metronomic chemotherapy in patients with T2 and above and/or lymph node positive early triple negative breast cancer who still had invasive tumor after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients with triple negative breast cancer diagnosed by biopsy in Peking University People's Hospital;
* 2) The clinical stages before treatment were T1-T4, N0-N3, M0;
* 3) Received treatment and operation in our hospital, and had hospitalization records;
* 4) Neoadjuvant chemotherapy is unlimited, and immunotherapy is allowed in neoadjuvant and/or adjuvant treatment;
* 5) Postoperative pathology confirmed the presence of residual invasive breast cancer in the breast and/or axillary lymph nodes;
* 6) Has signed and agreed to participate in the PKUPH breast disease cohort study.

Exclusion Criteria:

* 1) Lack of clinical and pathological data (such as imaging data and pathological data);
* 2) Patients with metastatic breast cancer or bilateral breast cancer;
* 3) Failure to perform radical surgery;
* 4) BRCA has pathogenic or possibly pathogenic mutations, and received intensive treatment with PARP inhibitors after operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Triple negative patients, non-PCR after neoadjuvant therapy
Sampling Method: Probability Sample
Enrollment: 1166 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure, including ipsilateral local recurrence, contralateral breast cancer, distant recurrence or death from any cause.

SECONDARY OUTCOMES:
invasive disease free survival | 5 years
  The time from study enrollment to the first occurrence of the following events defined as failure: local recurrence of ipsilateral invasive breast cancer, contralateral invasive breast cancer, distant recurrence or death from any cause.
distant disease free survival | 5 years
  Time from study enrollment to distant recurrence and metastasis
breast cancer specific survival | 5 years
  Time from study enrollment to death due to breast cancer
overall survival | 5 years
  Time from study enrollment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China